CLINICAL TRIAL: NCT02386215
Title: The Use of HIV Self-tests to Promote Partner and Couples Testing: a Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Impact Research & Development Organization (Other)
Responsible Party: Principal Investigator, Harsha Thirumurthy, PhD, Associate Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 14-3040
Record Dates: First submitted 2015-03-05; First posted 2015-03-11 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: HIV
Keywords: HIV self-testing; randomized controlled trial; Kenya

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIV Self-test (Experimental): Following a baseline interview, participants in the intervention group will be shown how to correctly use the self-tests and given two HIV self-tests. Subsequently, we will contact participants periodically over a 3 month period to see if they have used the test(s) with their sexual partners and conduct a follow-up interview.
  Interventions: Behavioral: HIV self-test
- Control (No Intervention): Following the baseline interview, participants in the control group will be given referral vouchers for themselves and their partners to obtain HIV testing at Voluntary Counseling & Testing (VCT) centers. We will contact the participants at the end of 3 months to see if they and/or their partner(s) have sought HIV testing.

INTERVENTIONS:
Behavioral: HIV self-test — Two self-test kits will be distributed to women, each containing the following:
  * One standard OraQuick ADVANCE I/II test kit
  * Written pre-test information including test instructions in written and pictorial form
  * A phone number that participants can call to obtain additional information
  * Two vouchers with unique identifying numbers which can be redeemed at confirmatory testing
  Other Names: Oraquick
  Arms: HIV Self-test

SUMMARY:
This randomized controlled trial will explore whether the provision of oral HIV self-test kits to women can increase HIV testing among their male partners. The study will recruit adult women from antenatal care and post-partum clinics in Kisumu. Each participant will be randomized to either receive two HIV self-tests or to receive counseling referring their partner to HIV testing (standard of care). Over a 3 month period, we will obtain information from study participants on how many sexual partners they offered the tests to, the receptivity of their sexual partners to using self-tests, and the incidence of any adverse events. We will compare partner testing rates in intervention and control groups.

DETAILED DESCRIPTION:
This randomized controlled trial will enroll women, ages 18-39, attending antenatal care (ANC) and post-partum care (PPC) at 3 sites in Kisumu, Kenya. The study's purpose is to investigate whether offering multiple HIV self-tests to women can increase the likelihood that either partner or couples HIV testing takes place.

Women who are randomized to the intervention group will be provided with multiple oral self-tests as well as information about how to use the tests and where to seek care if necessary. These women will be encouraged to give the self-tests to their sexual partners and encourage those partners to take a self-test. Women who are randomized to the control group will be offered the standard counseling to refer their partners for clinic-based HIV counseling and testing. Our hypothesis is that the intervention group will have higher uptake of HIV testing by women's partners within 3 months of enrollment in the study than the control group. Participants in the study will complete a baseline interview and a follow-up interview at 3 months post-enrollment. Qualitative in-depth interviews will be conducted with a subset of participants in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Primarily resides in or near Kisumu
* Reports having a current, primary partner (someone that the woman has been in a relationship with for at least 6 months and is identified as her primary partner)
* Reports that primary partner has not tested for HIV in past 6 months
* Have undergone the opt-out HIV testing at the ANC or PPC clinic
* Intends to continue living in or around Kisumu for the next 3 months (follow-up period).

Exclusion Criteria:

* Believes that her partner will hurt her if she gives him an HIV self-test and encourages him to use it
* Reports having an HIV+ partner
* Intends to relocate from Kisumu area within the next 3 months

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Proportion of partners that uptake HIV testing (questionnaire) | 3 months
  The primary outcome for the study will be uptake of HIV testing by women's partners within 3 months of enrollment in the study. For each participant, the investigators will record whether the participant's partner underwent HIV testing. The investigators will test for differences in the primary outcome variable between the intervention and control group.

SECONDARY OUTCOMES:
Proportion of participants who discussed HIV testing with partner (questionnaire) | 3 months
  Proportion of participants who report that they discussed HIV testing with their partner
Proportion of participants whose partners undergo HIV testing individually (questionnaire) | 3 months
  Proportion of participants whose partners undergo HIV testing individually (partner testing)
Proportion of participants who undergo Couples HIV testing with their partners (questionnaire) | 3 months
  Proportion of participants who undergo HIV testing with their partners (Couples testing)

CONTACTS AND LOCATIONS:
Overall Officials: Harsha Thirumurthy, PhD, Principal Investigator — University of North Carolina, Chapel Hill

REFERENCES:
- [Derived] Masters SH, Agot K, Obonyo B, Napierala Mavedzenge S, Maman S, Thirumurthy H. Promoting Partner Testing and Couples Testing through Secondary Distribution of HIV Self-Tests: A Randomized Clinical Trial. PLoS Med. 2016 Nov 8;13(11):e1002166. doi: 10.1371/journal.pmed.1002166. eCollection 2016 Nov. PMID 27824882